CLINICAL TRIAL: NCT02040207
Title: AM-101 in the Post-Acute Treatment of Peripheral Tinnitus 2 (AMPACT2) - an Open-Label Extension to the TACTT3 Study
Brief Title: AM-101 in the Treatment of Post-Acute Tinnitus 2
Acronym: AMPACT2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Auris Medical AG (Industry)
Responsible Party: Sponsor
Organization: Auris Medical, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AM-101-CL-12-04
Record Dates: First submitted 2014-01-14; First posted 2014-01-20 (Estimated); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — PDCD5 protein, rat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AM-101 injection (Experimental): AM-101 gel for intratympanic injection
  Interventions: Drug: AM-101

INTERVENTIONS:
Drug: AM-101 — AM-101 gel for intratympanic injection

SUMMARY:
The purpose of this research study is to test the safety and local tolerance of repeated treatment with AM-101.

DETAILED DESCRIPTION:
This open-label extension study is assessing the safety and local tolerance of repeated treatment with AM-101 in subjects previously treated in the scope of the TACTT3 study.

ELIGIBILITY:
Inclusion Criteria:

* Completion of TACTT3 study;
* Negative pregnancy test (woman of childbearing potential);
* Willing and able to attend the study visits.

Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Adverse event leading to treatment discontinuation in TACTT3;
* Meniere's Disease, endolymphatic hydrops, acoustic neuroma, severe or fluctuating hearing loss, otitis media, otitis externa, abnormality of tympanic membrane;
* Ongoing drug-based therapy for otitis media or otitis externa;
* Drug-based therapy known as potentially tinnitus-inducing;
* Other treatment of tinnitus;
* Drug abuse or alcoholism;
* Subjects with psychiatric diseases requiring drug treatment;
* Use of antidepressant or anti-anxiety medication;
* Any clinically relevant disorder or abnormality in physical examination;
* Women who are breast-feeding, pregnant or who are planning to become pregnant during the study;
* Women of childbearing potential who are unwilling or unable to practice contraception.

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 487 (Actual)
Dates: Start 2014-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Hearing threshold | Up to Day 203
  Occurrence of deterioration in hearing threshold in the treated ear(s)

SECONDARY OUTCOMES:
Hearing threshold | Up to Day 252
  Difference and occurence of deterioration of hearing threshold in the treated ear(s)
Adverse events and serious adverse events | Up to Day 252
  Occurrence and severity of adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational site, Munich, Germany

REFERENCES:
- See also: Link to Result entry in clinicaltrialsregister.eu — https://www.clinicaltrialsregister.eu/ctr-search/trial/2013-001527-39/results